CLINICAL TRIAL: NCT00432614
Title: A Multi-National, Multi-Center, DB, Placebo-Controlled, Parallel Group, Fixed Dose Efficacy & Safety Study of SR58611A 350 mg Twice Daily vs. Placebo in Adults With Major Depressive Disorder on Concomitant Treatment With Escitalopram 10mg/d
Brief Title: Efficacy and Safety of SR58611A co-Administered With Escitalopram in Adults With Major Depressive Disorder
Acronym: ALBERIO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC6224; EudraCT 2006-004146-16
Record Dates: First submitted 2007-02-07; First posted 2007-02-08 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Major Depressive Disorder
Keywords: Mental Disorder; Mood Disorder; Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Mental Disorders; Mood Disorders; Depressive Disorder | interventions — Amibegron hydrochloride; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Group 1 (Experimental): SR58611A 350mg twice daily with escitalopram 10mg once daily
  Interventions: Drug: SR58611A; Drug: escitalopram
- Group 2 (Active Comparator): placebo with escitalopram 10mg once daily
  Interventions: Drug: escitalopram
- Group 3 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SR58611A — oral administration
  Arms: Group 1
Drug: escitalopram — oral administration
  Arms: Group 1; Group 2
Drug: placebo — oral administration
  Arms: Group 3

SUMMARY:
The primary objective of the study is to compare, after 8 weeks, the efficacy of SR58611A vs. placebo in patients with Major Depressive Disorder who are on concomitant treatment with escitalopram.

The secondary objective of this study is to document clinical safety and tolerability of SR58611A in association with escitalopram.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients or outpatients with Major Depressive Disorder characterized by a recurrent Major Depressive Episode with Montgomery and Asberg Depression Rating Scale (MADRS) total score => 30

Exclusion Criteria:

* Patient is at immediate risk for suicidal behavior
* Patient with psychotic features, catatonic features, seasonal pattern or postpartum onset
* Patients with a current depressive episode secondary to a general medical disorder
* Patients with a lifetime history or presence of bipolar disorder, psychotic disorder, panic disorder and antisocial personality disorder
* Patients with severe or unstable concomitant medical conditions
* Pregnant, breastfeeding, or likely to become pregnant during the study
* Treated with escitalopram within 6 months before the study, or who have had an adverse reaction to escitalopram

The investigator will evaluate whether there are other reasons why a patient may not participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Hamilton Depression Rating scale (HAM-D) total score | 8 weeks

SECONDARY OUTCOMES:
Speed of response based on HAM-D and change in Clinical Global Impression (CGI) severity score | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (13):
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Tatari, Estonia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, Casablanca, Morocco
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)